CLINICAL TRIAL: NCT04726280
Title: Respiratory Impact of Local Anaesthetic Volume for an Interscalene Brachial Plexus Block With an Extrafascial Approach.
Brief Title: Respiratory Impact of LA Volume After IS Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eric Albrecht (Other)
Responsible Party: Sponsor-Investigator, Eric Albrecht, Sponsor-Investigator, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-02930
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Arthroscopic Surgery of the Shoulder; Extrafascial Interscalene Plexus Brachial Block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 ml single-shot injection (Experimental): In the 10ml group, participants will have an interscalene brachial plexus with an extrafascial injection of 10 ml ropivacaine 0.75% at the level of C5-C6 nerves roots.
  Participants will also receive multimodal analgesia with injection of dexamethasone 8 mg iv, magnesium sulfate 40 mg kg^-1 iv, ketorolac 30 mg iv, and acetaminophen 1000 mg iv, according to the current practice in our institution.
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution
- 20 ml single-shot injection group (Active Comparator): In the 20ml group, participants will have an interscalene brachial plexus with an extrafascial injection of 20 ml ropivacaine 0.75% at the level of C5-C6 nerves roots.
  Participants will also receive multimodal analgesia with injection of dexamethasone 8 mg iv, magnesium sulfate 40 mg kg^-1 iv, ketorolac 30 mg iv, and acetaminophen 1000 mg iv, according to the current practice in our institution.
  Interventions: Drug: Ropivacaine 0.75% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.75% Injectable Solution — 10 ml extrafascial interscalene brachial plexus block
  Arms: 10 ml single-shot injection
Drug: Ropivacaine 0.75% Injectable Solution — 20 ml extrafascial interscalene brachial plexus block
  Arms: 20 ml single-shot injection group

SUMMARY:
The hypothesis of this study is that a reduced extrafascial volume of local anesthetic for an interscalene brachial plexus block is associated with a lower incidence of diaphragmatic hemiparalysis after an arthroscopic surgery of the shoulder, without any reduction of the analgesic efficacy.

DETAILED DESCRIPTION:
The hypothesis of this study is that a reduced extrafascial volume of local anesthetic for an interscalene brachial plexus block is associated with a lower incidence of diaphragmatic hemiparalysis after an arthroscopic surgery of the shoulder, without any reduction of the analgesic efficacy.

Our prospective randomized controlled trial will include two parallel groups: a group will receive a volume of 20 mls of ropivacaine 0.75%, while the other group will receive a volume of 10 mls.

All participants will have a preoperative ultrasound-guided interscalene brachial plexus with an extrafascial injection of 10 or 20 mls of ropivacaine 0.75%. In both groups, participants will have an examination of the hemidiaphgragm with the ultrasound, before and 30 min after the block. The respiratory function will also be assessed with a bedside spirometer before and after the block, and at 12 and 24 postoperative hours. During surgery all participants will receive multimodal analgesia inclusive of iv dexamethasone 8 mg, iv magnesium sulfate 40 milligram kg^2, iv ketorolac 30 milligrams, and iv acetaminophen 1000 milligrams, according to the current practice in our institution. In the postoperative period, Participants will be prescribed an IV pca of morphine.

Assignment to one of these two groups will be done according to a computer-generated list of random numbers, and the sealed envelopes method will be used.

ELIGIBILITY:
Inclusion Criteria:

* arthroscopic surgery of the shoulder
* ASA class 1 to 3
* age more than 18 years old

Exclusion Criteria:

* patient refusal or inability to understand and/or sign the inform consent
* contraindication for perineural block (allergy to local anesthetics, infection of puncture site, major coagulopathy, sensitive or motor deficiency on the operative side arm
* chronic alcool abuse
* opioid drug abuse or under substitution treatment
* patients known for allergies to paracetamol, non steroidal anti inflammatory drugs, dexamethasone, sulfate magnesium, ondansetron, droperidol, and omeprazole;
* patients under chronic corticotherapy
* patients known for malignant hyperthermia;
* patients with chronic kidney failure (Glomerular Filtration Rate < 20 ml/min)
* patients with severe pulmonary disease
* patients with history of neck surgery or radiotherapy on the operative side;
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence of hemidiaphragmatic paralysis | 30 minutes after the interscalene plexus brachial extrafascial injection

SECONDARY OUTCOMES:
Incidence of hemidiaphragmatic paralysis | at 2 and 24 postoperative hours
Presence of Dyspnea | in phase 1 recovery and at 12 and 24 postoperative
  Verbal question to the patient if he has dyspnea or not
Presence of PONV | in phase 1 recovery and at 12 and 24 postoperative
  Verbal question to the patient if he has dyspnea or not
Presence of Pruritus | in phase 1 recovery and at 12 and 24 postoperative hours
  Verbal question to the patient if he has pruritus or not
Presence of Claude-Bernard-Horner syndrome | in phase 1 recovery and at 12 and 24 postoperative hours
  Examination of the patient
Presence of Dysphonia | in phase 1 recovery and at 12 and 24 postoperative hours
  Verbal question to the patient if he has dysphonia or not
Forced expiratory volume in one second | 30 minutes after the interscalene plexus brachial extrafascial injection, and at 2, 12 and 24 postoperative hours
  in liters per second
Forced vital capacity | 30 minutes after the interscalene plexus brachial extrafascial injection, and at 2, 12 and 24 postoperative hours
  in liters
Peak expiratory flow | 30 minutes after the interscalene plexus brachial extrafascial injection, and at 2, 12 and 24 postoperative hours
  in liters per second
Installation time of sensory block | up to 30 minutes after the interscalene plexus brachial extrafascial injection
  in minutes
Installation time of motor block | up to 30 minutes after the interscalene plexus brachial extrafascial injection
  in minutes
Time to first dose of postoperative iv morphine | up to 24 hours postsurgery
  in hours
Pain scores at rest | in phase 1 recovery and at 12 and 24 postoperative hours
  Numeric pain intensity scale. Pain scores range from zero (no pain) to 10 (worst possible pain)
Pain scores on movement | in phase 1 recovery and at 12 and 24 postoperative hours
  Numeric pain intensity scale. Pain scores range from zero (no pain) to 10 (worst possible pain).
Cumulative postoperative iv morphine consumption | in phase 1 recovery and at 12 and 24 postoperative hours
  in milligrams
Duration of analgesic block | up to 24 hours postsurgery
  in minutes
Duration of motor block | up to 24 hours postsurgery
  in minutes
Duration of sensory block | up to 24 hours postsurgery
  in minutes
Satisfaction of the participants | at 24 postoperative hours
  Numeric satisfaction intensity scale. Satisfactions range from 0 (totally unsatisfied) to 10 (maximal satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV (Centre Hospitalier Universitaire Vaudois), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Renard Y, Grape S, Gonvers E, Rossel JB, Goetti P, Albrecht E. Respiratory impact of local anaesthetic volume after interscalene brachial plexus block with extrafascial injection: a randomised controlled double-blinded trial. Br J Anaesth. 2025 Apr;134(4):1153-1160. doi: 10.1016/j.bja.2024.12.010. Epub 2025 Jan 23. PMID 39855930